CLINICAL TRIAL: NCT06538610
Title: Feasibility Study of Ambulatory Holter Monitoring While Receiving Infusional Fluorouracil (5-FU) Chemotherapy
Brief Title: The 5-FU Holter Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Gut Cancer Foundation (Unknown); Auckland City Hospital (Other Government); The Heart Group (Unknown)
Responsible Party: Principal Investigator, Jane So, Principal Investigator, Auckland City Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTNZ-2022-08; U1111-1308-6717 (Other: The Universal Trial Number)
Record Dates: First submitted 2024-06-04; First posted 2024-08-06 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Gastrointestinal Malignancy
MeSH Terms: interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Holter monitor (Experimental): Holter monitor for 48 hours
  Interventions: Device: Holter monitor

INTERVENTIONS:
Device: Holter monitor — Holter monitor fitted from start of 5-FU infusion (Day 1) to 5-FU infusion ending (Day 3).
  Holter monitor to be worn for approximately 46-48 hours.

SUMMARY:
To assess the feasibility of using ambulatory ECG monitoring (Holter monitor) for patients receiving 5-FU chemotherapy

DETAILED DESCRIPTION:
5-fluorouracil (5-FU) is the key chemotherapy component in systemic treatment of colorectal cancer. However, 5-FU treatment is also associated with cardiotoxicity which can have devastating consequences.

Cardiotoxicity can be both symptomatic (e.g. chest pain, myocardial infarction (heart attack) and/or sudden death) as well as asymptomatic ('silent myocardial ischemia', which is only detectable by ECG). Data suggests that asymptomatic cardiotoxicity may be relatively common (~30% of patients).

About 69% of the cardiac events are seen during or within the first 72 hours of the first cycle of 5-FU.

The development of cardiotoxicity requires permanent discontinuation of 5-FU chemotherapy. There are no PHARMAC funded alternatives for patients who discontinue 5-FU due to cardiotoxicity. Discontinuation of 5-FU is likely to lead to a worse oncological outcome (survival time) for the patient.

One proposed mechanism for 5-FU cardiotoxicity involves fluoro-beta-alanine (FBAL), which is a metabolite formed when 5-FU is catalysed by the enzyme dihydropyrimidine dehydrogenase (DPD). The rationale for this feasibility study is to provide preliminary information required to develop a prospective pharmacokinetic study exploring plasma clearance of FBAL and 5-FU cardiotoxicity.

This study aims to determine i) whether the use of continuous ECG monitoring (ambulatory Holter monitoring) in real life conditions (over two days, while at home receiving infusional 5-FU chemotherapy), is able to appropriately assess these types of silent heart attacks (ST changes) and ii) the acceptability of this study to both patients and clinicians iii) the excretion rate of FBAL over the 48 hour time period & interpatient pharmacokinetic variability in FBAL excretion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of gastrointestinal malignancy
* Planned to receive either FOLFOX chemotherapy with any treatment intent
* Aged ≥ 18 years at time of signing informed consent form

Exclusion Criteria:

• ECG with left bundle branch block or left ventricular hypertrophy with strain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Up to 1 year
  The percentage of participants who were contacted and joined the study will be reported.
Acceptability rate | Up to 1 year
  The percentage of participants who joined the study and wore the Holter monitor for the required study duration.
Completion rate | Up to 1 year
  The percentage of participants who joined the study and completed all study assessments
Overall time required to recruit to the target sample size | Up to 1 year
  The overall time in weeks required to recruit participants for the feasibility study will be reported.
Clinician experience of recruitment | After 1 year
  Clinician Survey administered at end of study recruitment to measure clinicians' perceived ease of recruitment (5-point Likert scale 1=Difficult to 5=Very easy)
Clinician experience of barriers to recruitment | After 1 year
  Clinician Survey administered at end of study recruitment to measure clinicians' perceived barriers to recruitment (open ended questions)
Clinician experience of software module (Pathfinder SL) to measure ST segments using Holter monitoring while receiving infusional 5-FU chemotherapy | After 1 year
  Clinician Survey administered at the end of study recruitment to measure clinicians' perceived quality of Holter monitor recordings (5-point Likert scale 1=Poor to 5=Excellent)
FBAL (fluoro-beta-alanine) Excretion rate | 3 hours
  Cumulative urine sample collected over 3 hours
FBAL (fluoro-beta-alanine) Area under the Curve (AUC) | 0, 20 minutes, 1 hour, 3 hours
  Blood samples collected prechemo and 20 mins, 1 hour, 3 hours
FBAL (fluoro-beta-alanine) Clearance (CL) | 0, 20 minutes, 1 hour, 3 hours
  Blood samples collected prechemo and 20 mins, 1 hour, 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No